CLINICAL TRIAL: NCT01924013
Title: Randomized Placebo-controlled Trial of Maternal Vitamin D Supplementation During Pregnancy and Lactation to Improve Infant Linear Growth in Dhaka, Bangladesh.
Brief Title: Maternal Vitamin D for Infant Growth (MDIG) Trial
Acronym: MDIG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Shimantik (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Daniel Roth, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1000039072
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pregnancy
Keywords: Pregnancy; Infant Growth; Vitamin D; Bangladesh
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Placebo Comparator): Prenatal Period 0 IU; Postpartum Period 0 IU (placebo)
  Overall:The Prenatal Period will start at enrolment (17-24 weeks gestation) and last until delivery. The Postpartum Period will last from delivery until 6 months postpartum.
  Interventions: Dietary Supplement: Placebo
- Group B (Experimental): Prenatal Period 4,200 IU/week of vitamin D3 (=600 IU/d); Postpartum Period 0 IU/week (placebo)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol); Dietary Supplement: Placebo
- Group C (Experimental): Prenatal Period 16,800 IU/week of vitamin D3 (=2,400 IU/d); Postpartum Period 0 IU/week (placebo)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol); Dietary Supplement: Placebo
- Group D (Experimental): Prenatal Period 28,000 IU/week of vitamin D3 (=4,000 IU/d); Postpartum Period 0 IU/week (placebo)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol); Dietary Supplement: Placebo
- Group E (Experimental): Prenatal Period 28,000 IU/week of vitamin D3 (=4,000 IU/d); Postpartum Period 28,000 IU/week(=4,000 IU/d)
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol) — The intervention is an oral tablet containing vitamin D3 (cholecalciferol). This vitamin D supplement will be provided in the form of small tablets (approximately 10 mm diameter) and will be custom- manufactured by Toronto Institute for Pharmaceutical Technology (TIPT) in Toronto, Ontario, Canada. Each weekly dose will consist of a single tablet. Across trial groups, the tablets will only vary with respect to the vitamin D3 dose, as described above.
  Arms: Group B; Group C; Group D; Group E
Dietary Supplement: Placebo — This product will be identical in appearance, taste and texture to the experimental formulation but will not include any vitamin D3.
  Arms: Group A; Group B; Group C; Group D

SUMMARY:
The primary aims of this study are: 1) to determine whether maternal prenatal vitamin D3 supplementation (4200 IU/week, 16,800 IU/week, or 28,000 IU/week) versus placebo increases or decreases infant length at 1 year of age, and 2) to determine whether maternal postpartum vitamin D3 supplementation (28,000 IU/week) versus placebo increases or decreases length at 1 year of age among infants born to women who received vitamin D 28,000 U/week during pregnancy. Infants enrolled in the study will be followed for 2 years to document the persistence of any observed effects measured at 1 year of age. This study aims to enroll 1300 pregnant women in the 2nd trimester at a maternity hospital in Dhaka. Participants will be randomized to one of three doses of vitamin D3 (4200 IU/week, 16,800 IU/week, or 28,000 IU/week) or placebo throughout pregnancy. Women in the 28,000 IU/week group will be additionally randomized to either placebo or a continuation of 28,000 IU/week for 6 months postpartum. In addition to linear length, the trial will include analyses of inflammatory and hormonal determinants of infant growth, epigenetic phenomena that affect vitamin D metabolism, and diarrheal and respiratory morbidity in the infants.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and above.
* Gestational age of 17 to 24 completed weeks estimated based on recalled last menstrual period (LMP) and/or ultrasound.
* Intends to permanently reside in the trial catchment area for at least 18 months.

Exclusion Criteria:

* History of medical conditions that may predispose the participant to vitamin D sensitivity, altered vitamin D metabolism and/or hypercalcemia, or history of renal calculi.
* High-risk pregnancy based on one or more of the following findings by point-of-care testing:

  * Severe anemia: hemoglobin <70 g/L assessed by Hemocue
  * Moderate-severe proteinuria: ≥ 300 mg/dl (3+ or 4+) based on urine dipstick
  * Hypertension: systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg
* Multiple gestation, major congenital anomaly, or severe oligohydramnios based on maternal history and/or ultrasound.
* Unwillingness to stop taking non-study vitamin D or calcium supplements or a multivitamin with calcium and/or vitamin D.
* Currently prescribed vitamin D supplements as part of a physician's treatment plan for vitamin D deficiency.
* Previous participation in the same study.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Infant Length-for-Age Z-Scores with Prenatal Supplementation | 1 year of age
Infant Length-for-Age Z-Scores with Postpartum Supplementation | 1 year of age
  A separate analysis will be performed to assess the effect of continuation of 28,000 IU/week postpartum supplementation versus placebo (postpartum) among participants randomized to 28,000 IU/week prenatal.

SECONDARY OUTCOMES:
Serum calcium | 17 weeks gestation to birth (prenatal) and over 2 years postpartum
  Maternal serum calcium will be measured during pregnancy as a primary biochemical safety parameter and post partum.

OTHER OUTCOMES:
Stunting (LAZ < -2 SD below the median) at 1 and 2 years of age. | 1-2 years
Attained length and LAZ at 2 years of age. | 2 years postnatal
Birth weight, low birth weight %, small-for-gestational age % | Birth
Preterm birth % | Birth
Stillbirth % | 17 weeks gestation to 39 weeks
  Prenatal period
Maternal, perinatal, neonatal and infant severe morbidity and mortality | From 17 weeks gestation to 6 months postpartum
  During intervention phase (prenatal and first 6 months postpartum)
Infant acute respiratory infections and diarrhea | 6 months postpartum
  first 6 months postnatal
Biomarker concentrations (specific hormones, nutrients, environmental contaminants, and inflammatory markers potentially involved in the mediation or modification of the effect of vitamin D on infant stunting). | 17 weeks gestation to 2 years postpartum
  Prenatal and first 2 years postnatal
Epigenetic patterns of genes involved in vitamin D metabolism. | Birth

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Palacios C, Kostiuk LL, Cuthbert A, Weeks J. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2024 Jul 30;7(7):CD008873. doi: 10.1002/14651858.CD008873.pub5. PMID 39077939
- [Derived] Pell LG, Ohuma EO, Yonemitsu C, Loutet MG, Ahmed T, Mahmud AA, Azad MB, Bode L, Roth DE. The Human-Milk Oligosaccharide Profile of Lactating Women in Dhaka, Bangladesh. Curr Dev Nutr. 2021 Nov 13;5(12):nzab137. doi: 10.1093/cdn/nzab137. eCollection 2021 Dec. PMID 34993388
- [Derived] O'Callaghan KM, Shanta SS, Fariha F, Harrington J, Mahmud AA, Emdin AL, Gernand AD, Ahmed T, Abrams SA, Moore DR, Roth DE. Effect of maternal prenatal and postpartum vitamin D supplementation on offspring bone mass and muscle strength in early childhood: follow-up of a randomized controlled trial. Am J Clin Nutr. 2022 Mar 4;115(3):770-780. doi: 10.1093/ajcn/nqab396. PMID 34849536
- [Derived] Jukic AMZ, Zuchniak A, Qamar H, Ahmed T, Mahmud AA, Roth DE. Vitamin D Treatment during Pregnancy and Maternal and Neonatal Cord Blood Metal Concentrations at Delivery: Results of a Randomized Controlled Trial in Bangladesh. Environ Health Perspect. 2020 Nov;128(11):117007. doi: 10.1289/EHP7265. Epub 2020 Nov 23. PMID 33226277
- [Derived] Subramanian A, Korsiak J, Murphy KE, Al Mahmud A, Roth DE, Gernand AD. Effect of vitamin D supplementation during pregnancy on mid-to-late gestational blood pressure in a randomized controlled trial in Bangladesh. J Hypertens. 2021 Jan;39(1):135-142. doi: 10.1097/HJH.0000000000002609. PMID 32773651
- [Derived] Jeong JH, Korsiak J, Papp E, Shi J, Gernand AD, Al Mahmud A, Roth DE. Determinants of Vitamin D Status of Women of Reproductive Age in Dhaka, Bangladesh: Insights from Husband-Wife Comparisons. Curr Dev Nutr. 2019 Oct 7;3(11):nzz112. doi: 10.1093/cdn/nzz112. eCollection 2019 Nov. PMID 31723723
- [Derived] Roth DE, Morris SK, Zlotkin S, Gernand AD, Ahmed T, Shanta SS, Papp E, Korsiak J, Shi J, Islam MM, Jahan I, Keya FK, Willan AR, Weksberg R, Mohsin M, Rahman QS, Shah PS, Murphy KE, Stimec J, Pell LG, Qamar H, Al Mahmud A. Vitamin D Supplementation in Pregnancy and Lactation and Infant Growth. N Engl J Med. 2018 Aug 9;379(6):535-546. doi: 10.1056/NEJMoa1800927. PMID 30089075
- [Derived] Roth DE, Gernand AD, Morris SK, Pezzack B, Islam MM, Dimitris MC, Shanta SS, Zlotkin SH, Willan AR, Ahmed T, Shah PS, Murphy KE, Weksberg R, Choufani S, Shah R, Al Mahmud A. Maternal vitamin D supplementation during pregnancy and lactation to promote infant growth in Dhaka, Bangladesh (MDIG trial): study protocol for a randomized controlled trial. Trials. 2015 Jul 14;16:300. doi: 10.1186/s13063-015-0825-8. PMID 26169781